CLINICAL TRIAL: NCT06858189
Title: Can Nature-based Physical Activity Improve Symptoms of Depression and Anxiety?
Brief Title: Promoting Active Therapy: Path to Wellness
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kansas State University (Other)
Collaborators: REI Cooperative Action Fund (Unknown)
Responsible Party: Principal Investigator, Emily Mailey, Associate Professor, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB12197
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Depression, Anxiety; Physical Activity; Time in Nature; Self-Efficacy; Feasibility Pilot Study
Keywords: therapy; nature prescriptions; park prescriptions (ParkRx); exercise; mental health; walk-and-talk
MeSH Terms: conditions — Depression; Anxiety Disorders; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (immediate start) (Experimental): Participants will engage in walk-and-talk therapy during weekly sessions with their therapist and will set goals for engaging in nature-based physical activity on their own outside of therapy.
  Interventions: Behavioral: Walk-and-talk therapy
- Waitlist control (No Intervention): Participants will receive generic educational materials about nature-based physical activity and local parks.

INTERVENTIONS:
Behavioral: Walk-and-talk therapy — During the 10-week intervention, clients and therapists will engage in walk-and-talk therapy outdoors in natural settings during weekly therapy sessions. In addition, therapists will work with clients to set realistic goals for increased nature-based physical activity outside of the therapy setting. Therapists will check in with clients weekly regarding their progress and assist with goal revision, barrier planning, and self-monitoring.
  Other Names: Path to Wellness
  Arms: Intervention (immediate start)

SUMMARY:
This project will examine changes in depression and anxiety following a 10-week intervention promoting nature-based physical activity in mental health settings. We will recruit ten licensed therapists whose caseload includes adults with depression and anxiety. Following a training by our team, each participating therapist will recruit six clients, who will be randomly assigned to the intervention or control condition. Clients in the intervention condition will engage in walk-and-talk therapy outdoors during weekly sessions and discuss strategies for being active outdoors on their own. We will assess changes in depression, anxiety, and nature-based physical activity in both groups.

DETAILED DESCRIPTION:
For this project, we will recruit ten licensed therapists whose caseload includes adults with depression and anxiety. We aim to recruit therapists who practice in northeast Kansas. Our team will lead a 3-hour in-person training for participating therapists that covers project aims and procedures, benefits of nature-based physical activity for mental health, identifying and enrolling suitable clients for participation, recommending and engaging in nature-based physical activity with clients, and completing project assessments.

Following the training, each therapist will recruit six clients aged 18-65 who are willing to participate in a 10-week research study and meet the following criteria: 1) diagnosed depressive or anxiety disorder, 2) able to safely engage in moderate physical activity, and 3) willing to complete all research requirements. Clients who are part of an underrepresented minority group (i.e., racial/ethnic minority, low SES, LGTBQ) will be prioritize during recruitment. Therapists will invite eligible clients to participate in the study, and those who agree will sign an informed consent document. Clients will be randomly assigned to the intervention or active waitlist control (usual care) condition. All participants will receive a Fitbit and download the NatureDose app. During the 10-week intervention, clients and therapists will engage in walk-and-talk therapy outdoors in natural settings during weekly therapy sessions. In addition, therapists will work with clients to set realistic goals for increased nature-based physical activity outside of the therapy setting. Therapists will check in with clients weekly regarding their progress and assist with goal revision, barrier planning, and self-monitoring. Control participants will receive information about nature-based physical activity, and then will receive the full intervention after 10 weeks.

All participating clients will complete surveys assessing depression and anxiety symptoms at baseline (following informed consent) and at the end of the 10-week intervention. Throughout the 10-week intervention, therapists will keep a weekly log of frequency and duration of walk-and talk sessions. Clients will also keep a weekly log of nature-based physical activity, use the NatureDose app to measure time spent in nature each day, and wear a Fitbit to track their daily physical activity. At the end of the intervention, clients will complete a brief satisfaction survey, and therapists will complete an individual interview with the research team.

ELIGIBILITY:
Inclusion Criteria:

* Current client of a participating therapist who has completed study training
* Diagnosed depressive or anxiety disorder
* Able to safely engage in moderate physical activity
* Willing to complete all study requirements

Exclusion Criteria:

* Planning to discontinue therapy in less than 6 months
* Active suicidal ideation
* Does not pass exercise risk screener

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Participation in walk-and-talk therapy | Weekly throughout the 10-week intervention
  Therapists will keep logs of weekly attendance and participation in walk-and-talk therapy during sessions. Outcome will be calculated as a percentage of offered sessions.
Perceived therapist support for nature-based physical activity | End of intervention (after 10 weeks)
  Participating clients will complete a survey indicating how frequently their therapist asks about physical activity, recommends physical activity, engages in physical activity with the client, etc.
Acceptability | End of intervention (after 10 weeks)
  At the end of the intervention, clients will complete a survey indicating how much the discussions/sessions were helpful, enjoyable, informative, etc.

SECONDARY OUTCOMES:
Self-efficacy for physical activity | baseline, 10 weeks
  Measured with a modified version of the barriers self-efficacy scale
Self-efficacy for time in nature | baseline, 10 weeks
  Measured with the self-efficacy for spending time in nature scale
Physical activity | Weekly throughout the 10-week intervention
  Average MVPA and daily steps measured via Fitbit inspire 3 devices
Time in nature | Weekly throughout the 10-week intervention
  Measured via NatureDose app

OTHER OUTCOMES:
Depression | baseline, 10 weeks
  Measured via PHQ-9
Anxiety | baseline, 10 weeks
  Measured via GAD-7

CONTACTS AND LOCATIONS:
Locations (1):
- Kansas State University, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided